CLINICAL TRIAL: NCT06940674
Title: Adjunctive Cannabidiol for Recovery From Opioid Study (ACROS)
Brief Title: Adjunctive Cannabidiol for Recovery From Opioid Study
Acronym: ACROS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); International Center for Health Outcomes and Innovation Research (Other); Brains Bioceutical (Unknown)
Responsible Party: Principal Investigator, Yasmin Hurd, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-24-01494; UH3DA050323 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder (OUD)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Randomization will be carried out within each site using stratification factors. Using stratified block randomization with randomly varying block sizes, participants who meet the eligibility requirements and provide informed consent will be randomly allocated to one of the study arms (1 capsule CBD (200 mg), 2 capsules CBD (400 mg), 1 capsule placebo and 2 capsules placebo) with a 1:1:0.5:0.5 allocation ratio. The placebo groups will be combined for statistical analysis purposes. Random permuted blocks sizes within stratification groups will be used to minimize the chance of selection bias.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators and participants will be blinded to treatment assignment. The staff involved in primary outcome assessment and laboratory tests in local laboratories will also be blinded to treatment assignment. Randomization will be generated centrally and performed through a Web-based data collection system that automates the delivery of the randomization codes. The treatment assignment will be sent to the unblinded pharmacist or unblinded study team electronically, in a secure fashion, and electronic verification of the treatment assignment will be required before proceeding with the treatment intervention. Active drug and placebo will be identical to maintain study blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 capsule CBD (200 mg) (Experimental): 1 capsule 200 mg CBD 2x per day
  Interventions: Drug: Cannabidiol
- 2 capsules CBD (400 mg) (Experimental): 2 capsules 400 mg CBD 2x per day
  Interventions: Drug: Cannabidiol
- 1 capsule placebo and 2 capsules placebo (Placebo Comparator): 1 capsule 200 mg placebo 2x per day or 2 capsules 400 mg placebo 2x per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — 1 capsule CBD 200mg
  Other Names: CBD
  Arms: 1 capsule CBD (200 mg); 2 capsules CBD (400 mg)
Drug: Placebo — Bovine Gel Placebo capsule
  Arms: 1 capsule placebo and 2 capsules placebo

SUMMARY:
The long-term goal of the project is to determine whether cannabidiol (CBD) can reduce craving and relapse in individuals with opioid use disorder (OUD). The first phase of this project was an open cross-over design study in healthy individuals to confirm the safety and pharmacokinetic (PK) effects of CBD (BSPG CBD; Brains Bioceutical). The second phase was a double-blinded randomized controlled trial to determine whether CBD reduces craving and anxiety in individuals with OUD maintained on opioid agonist therapy. This phase 3 trial will determine whether CBD can serve as a potential adjunct treatment to reduce illicit opioid use in individuals with OUD maintained on opioid agonist therapy.

DETAILED DESCRIPTION:
Responding to the urgent calls for developing non-opioid therapeutics to address the opioid addiction epidemic, we have been investigating the therapeutic potential of cannabidiol (CBD), a non-intoxicating cannabinoid as a possible strategy. Our preclinical animal studies demonstrated that CBD decreases cue-induced heroin seeking behavior during drug abstinence, associated with the incubation of craving. Moreover, the effects of CBD to reduce heroin-seeking behavior was still evident even in animals that were maintained on methadone. We also showed in randomized, double-blind placebo- controlled design human clinical trials that acute CBD (Epidiolex) administration (400 mg and 800mg) decreased craving and anxiety associated with heroin cues in abstinent individuals with heroin use disorder, an effect that persisted even a week after the last CBD dose (given daily for 3 days). Moreover, another of our human studies showed that CBD was safe even in combination with a potent opioid agonist (fentanyl) to address a potential relapse condition suggesting negligible negative interaction with opioids. Building on those studies, we next set out to investigate the potential for CBD as an adjunctive treatment to methadone or buprenorphine in opioid use disorder (OUD). To that end, we first conducted Phase 1 pharmacokinetic studies with a CBD formulation in oral capsules (BSPG CBD; Brains Bioceutical) in healthy participants that showed that oral administration of BSPG CBD (400 mg) led to comparable pharmacokinetic parameters of the CBD plasma levels and its active metabolite as Epidiolex (400 mg), an FDA-approved comparator CBD product that previously reduced craving. In the Phase 2 clinical trial, we evaluated the effect of 200mg CBD (vs placebo) twice daily for 4 weeks and an additional 4 weeks of 400 mg CBD, twice daily, on cue-induced craving and anxiety in individuals with OUD who are maintained on methadone or buprenorphine. In the next phase of this IND application, we will extend the Phase 2 study to evaluate the effects of 200mg CBD, 400 mg CBD and placebo, taken twice daily, over a 24-week period in the OUD individuals maintained on methadone or buprenorphine. Our goals in this double-blinded randomized controlled clinical trial (RCT) are to investigate the potential of CBD to 1) decrease illicit opioid use and 2) reduce craving.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 65 years old.
* Ability to understand and give informed consent.
* Current opioid use disorder (OUD) or OUD in remission while on maintenance therapy with OAT, as determined by DSM-5 with the M.I.N.I. interview (Mini-International Neuropsychiatric Interview).
* Current opioid agonist maintenance treatment with methadone or buprenorphine for at least 14 days prior to consent. With the following more specific criteria for each of these two medications:

  * Current methadone maintenance treatment with a dose of ≥ 10mg/day, (maximum: 250mg/day), AND urinary toxicology positive for methadone and 2-ethylidene-1,5-dimethyl-3,3-diphenylpyrrolidine (EDDP).
  * Current buprenorphine maintenance treatment with a dose of ≥ 2mg/day (maximum: 32mg/day), AND urinary toxicology positive for buprenorphine.

Exclusion Criteria:

* Participants who are non-English speaking.
* Psychiatric conditions under DSM-5 (examined with the MINI) that would make study participation unsafe, or which would prevent adherence to study procedure; examples include: suicidal (i.e. high risk for suicide on the Columbia suicide severity rating scale (C-SSRS) screen version) or homicidal ideation requiring immediate attention, inadequately-treated mental health disorder (e.g., active psychosis, uncontrolled bipolar disorder).
* Current diagnosis of a severe substance use disorder (except for opioid and nicotine/tobacco) in the past 3 months, based on the MINI interview, that would preclude safe participation in the study as determined by the study medical clinician.
* Signs of acute drug intoxication when arriving at the study site as determined by clinician assessment.
* Medical or psychiatric contraindications for CBD administration (e.g., history of hypersensitivity to cannabinoids); or any of the ingredients in the product (gelatin or sesame oil).
* Showing signs of acute opioid withdrawal symptoms (as determined by the result of the Clinical Opiate Withdrawal Scale (COWS). A Score of ≥ 5 or as interpreted by the investigator will be considered a positive result for withdrawal symptoms).
* Have a medical condition that would make study participation unsafe, which would make treatment compliance difficult, or would prevent adherence to study procedure. This includes but is not limited to the following criteria: • < 30mL/min/1.73m2 eGFR. •QTc Fridericia > 500ms at screening. •Elevated liver enzymes at screening. The exclusionary lab values are: >4x the upper limit of normal (ULN) per laboratory criteria for AST or ALT or >1.5x ULN for bilirubin.
* Participating in another pharmacotherapeutic trial in the past 3 months.
* Participants who have used (within 14 days prior to consent) or plan to use (during the 24-week treatment period) any medications, dietary supplements (and/or grapefruit juice), or combination of medications and supplements known to alter the metabolism of, or interact with CBD (buproprion, rifampin, barbiturates, phenothiazines, cimetidine, anticoagulants, antiplatelets, etc.).
* For women: being pregnant (positive urine test for pregnancy) or breastfeeding.
* Not using an appropriate method of contraception such as hormonal contraception (oral hormonal contraceptives, Depo-Provera, Nuva-Ring), intrauterine device (IUD), sterilization, or double barrier method (combination of any two barrier methods used simultaneously, i.e. condom, spermicide, diaphragm).
* Participants who have been court mandated to attend treatment centers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of study participants with negative urine toxicology for illicit opioid use | 24 weeks
  Percentage of study participants with negative urine toxicology for illicit opioid use over the course of 24 weeks.

SECONDARY OUTCOMES:
Concentration of illicit opioids | Duration of the trial, 24 weeks
  Concentration of illicit opioids in quantitative plasma toxicology (plasma every four weeks)
Weeks of abstinence | Duration of the trial, 24 weeks
  Weeks of abstinence of illicit opioid use
Use of non-opioid illicit substances | Duration of the trial, 24 weeks
  Number of weeks using other non-opioid illicit substances
Duration of first opioid abstinence | Duration of the trial, 24 weeks
  Duration of first opioid abstinence, defined as the number of weeks from randomization to first opioid test positive or urine test missed.
Cue-induced Visual Analog Scale for craving (VASC) | At 12 and 24-week time points
  Cue-induced Visual Analog Scale for craving (VASC)
  Cue-induced Visual Analog Scale for craving is used to measure subjective craving responses to a drug and neutral video cues evaluated in the clinic. Total scale ranges from 0-10, with higher scores indicating extreme cravings.
Cue-induced Visual Analog Scale for anxiety (VASA) | At 12 and 24-week time points
  Cue-induced Visual Analog Scale for anxiety (VASA)
  Cue-induced Visual Analog Scale Anxiety is used to measure subjective anxiety responses to a drug and neutral video cue evaluated in the clinic. Total scale from 0-10, with higher score indicating extreme anxiety.
Change in illicit opioids in plasma toxicology | 24 weeks
  Change in illicit opioids in plasma toxicology
Change in illicit opioids in urine toxicology | 24 weeks
  Change in illicit opioids in urine toxicology
Study Retention | 24 weeks
  Number of participants remaining in the study
Opioid Craving Questionnaire (OCQ) | Every 4 weeks up to 24 weeks
  General craving self-report using Opioid Craving Questionnaire (OCQ)
  Total scale from 0-9, with higher score indicating more severe craving
Generalized Anxiety Disorder Scale (GAD7) | Every 4 weeks up to 24 weeks
  General anxiety self-report using the Generalized Anxiety Disorder Scale (GAD7).
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms.
Substance use other than opioids | Duration of the trial, 24 weeks
  Proportion of substance use other than opioids
Methadone plasma concentrations | Duration of the trial, 24 weeks
  Methadone plasma concentrations
Buprenorphine and metabolite plasma concentrations | Duration of the trial, 24 weeks
  Buprenorphine and metabolite plasma concentrations
Retention in opioid agonist therapy | Duration of the trial, 24 weeks
  Proportion of participants who remained in treatment with opioid agonist therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hurd, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - CODA Treatment Recovery, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Data will be shared no later than 6 months after study completion or as soon as any necessary cleaning and validation procedures are performed.
Access Criteria: There are no major factors affecting the access, distribution or reuse of the scientific data to be generated. All research participants will be consented for broad data sharing. All data will be made publicly available once the study is completed, following the timeline outlined in Element 4. The data will be de-identified to ensure study participant confidentiality. Access to the scientific data will not be controlled other than the requirements imposed by the NDA and IRB as mentioned above. Data will be distributed via publicly accessible platforms, including the HEAL Data Commons and ClinicalTrials.gov. These repositories ensure that the data is accessible to the broader scientific community. Data reuse will be encouraged as long as it adheres to the HEAL Data Commons' data use and citation policies as well as any requirements imposed by the IRB. Data users must acknowledge the original study and its investigators in any publications or other outputs based on the shared data.